CLINICAL TRIAL: NCT03816800
Title: Investigating the Association of Iron and Pollen Allergy in Female Subjects Studie Zur Wirkung Von Eisen Auf Pollenallergikerinnen
Brief Title: Iron and Pollen Allergy in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Franziska Roth-Walter, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1370/2018
Record Dates: First submitted 2019-01-21; First posted 2019-01-25 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Allergy Pollen; Healthy
Keywords: Allergy; iron-deficiency; birch; grass
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Hypersensitivity; Anemia, Iron-Deficiency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-Allergic (Placebo Comparator): Over the course of 6 months allergic participants receive twice daily a placebo tablets.
  Interventions: Dietary Supplement: Placebo
- Active-Allergic (Active Comparator): Over the course of 6 months allergic participants receive twice daily a dietary supplement containing whey protein-bound, chelated iron.
  Interventions: Dietary Supplement: ImmunoBon

INTERVENTIONS:
Dietary Supplement: ImmunoBon — The dietary agent contains vitamin A, Zn, chelated iron and whey proteins.
  Arms: Active-Allergic
Dietary Supplement: Placebo — the dietary agent does not contain vitamin A, Zn, chelated iron and whey proteins
  Arms: Placebo-Allergic

SUMMARY:
Iron deficiency and anemia are clearly associated with the onset of allergy and allergic diseases, whereas an improved iron status seems to prevent the onset of allergy in humans. Iron-deficiency can be absolute or functional. Functional iron-deficiency occurs during immune activation and may be reflective for the hyperactive state of atopic subjects.

The investigators plan a prophylactic dietary intervention study in atopic/allergic and non-allergic individuals that transport chelated iron to immune cells. Over the course of six months, oral supplementation of placebo or whey protein-bound chelated iron will be given and 1) clinical reactivity 2) iron status and 3) changes in the microflora due to the treatment will be assessed.

DETAILED DESCRIPTION:
There is no state-of-the-art prophylactic treatment for atopy. Once allergy develops, allergens should be avoided, and specific allergen immunotherapy applied. The initial cause of the onset of allergy, namely the immune hyperactive state of the atopic subjects, is not addressed at all. The investigators hypothesize that atopy is defined by a mild functional iron deficiency and that improving the iron status of immune cells will decrease the reactivity of these cells.

In this prophylactic dietary intervention study oral supplementation of placebo or chelated and whey protein-bound iron will be given over the course of six months to allergic and non-allergic women. Changes in 1) the clinical reactivity 2) the iron status and 3) the microflora will be assessed. The study will be the first systematic approach in humans to assess the contribution of iron deficiency to allergy and will be pivotal in supporting the implementation of prophylactic and therapeutic recommendations.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy premenopausal women over 18 years of age. Allergic participants should have been diagnosed with allergic rhinitis against birch and/or grass pollen.

Exclusion Criteria:

* Subjects with co-morbidities such as diabetes mellitus, disorders of the liver including hemochromatosis or kidney, autoimmune and metabolic diseases or malignancies or who use medications (e.g. antibiotics, PPIs) that influence the iron, inflammatory or microbial status will be excluded. Further exclusion criteria are pregnancy, lactation, zinc, and iron supplementation and smoking. Subjects with a history of major bleeding (including trauma, surgery, other major blood loss) within the last 2 years and blood transfusion within the last 2 years, or with a history of significant breakthrough bleeding will be excluded. Volunteers will be asked to cease blood donation at least three months before recruitment. Allergics with a history of an allergen-induced anaphylactic shock or with severe, uncontrolled asthma who in the last two years have received allergen immunotherapy or an anti-IgE therapy will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — premenopausal women
Enrollment: 58 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Symptom severity - Total nasal symptom score | Baseline
  Symptoms (with max 2 points for secretions, irritations and distant symptoms): score of 6 means all symptoms present (secretion, irritations and distant symptoms)
Symptom severity - Total nasal symptom score | 8 months
  Symptoms (with max 2 points for secretions, irritations and distant symptoms): score of 6 means all symptoms present (secretion, irritations and distant symptoms)

SECONDARY OUTCOMES:
Mean daily combined symptom medication score during the peak of the pollen season | up to 6 months
  The score will be recorded daily for 45-180 days during the pollen season
Iron status | Baseline
  Hemoglobin, Ferritin, hepcidin, hemopexin,ceruloplasmin, iron and soluble transferrin receptor concentrations, transferrin saturation in %
Iron status | 8 months
  Hemoglobin, Ferritin, hepcidin, hemopexin,ceruloplasmin, iron and soluble transferrin receptor concentrations, transferrin saturation in %
Exploratory - Microbiome | baseline
  microbial composition will be assessed by 16S rRNA sequencing in order to determine bacterial communities present in samples, their relative abundance and overall diversity. Samples: gastrointestinal and nasal samples
Exploratory - Microbiome | 8 months
  microbial composition will be assessed by 16S rRNA sequencing in order to determine bacterial communities present in samples, their relative abundance and overall diversity. Samples: gastrointestinal and nasal samples

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Roth-Walter, PhD, Principal Investigator — The interuniversity Messerli Research Institute
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Petje LM, Jensen SA, Szikora S, Sulzbacher M, Bartosik T, Pjevac P, Hausmann B, Hufnagl K, Untersmayr E, Fischer L, Vyskocil E, Eckl-Dorna J, Jensen-Jarolim E, Hofstetter G, Afify SM, Krenn CG, Roth GA, Rivelles E, Hann S, Roth-Walter F. Functional iron-deficiency in women with allergic rhinitis is associated with symptoms after nasal provocation and lack of iron-sequestering microbes. Allergy. 2021 Sep;76(9):2882-2886. doi: 10.1111/all.14960. Epub 2021 Jun 17. No abstract available. PMID 34037999